CLINICAL TRIAL: NCT04883931
Title: The Effect of Using Breast Milk as a Topical Ophthalmic Drop on Retinopathy of Prematurity. Randomized Placebo-controlled Trial.
Brief Title: Mother Milk as a Eye Drop & Premature Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Konya City Hospital (Other); Konya Dr. Ali Kemal Belviranli Hospital for Obstetrics and Pediatrics (Unknown)
Responsible Party: Principal Investigator, Musa Silahli, Principal Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KA21/65
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-05

CONDITIONS: Retinopathy of Prematurity
Keywords: Breast milk; Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Saline Solution; Milk, Human

STUDY DESIGN:
Intervention Model Description: Porspective Randomized Placebo Controlled Trail
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and Ophthalmologist who is the responsible the follow -up the ROP stages will be blind in the study. The neonatologist who is responsible for the care and follow-up of the patients will not be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): With in 48-72 hour after birth, infants will receive 0.5 ml breast milk for own mother as a eye drop twice in a day until the discharge or need for laser coagulation. Fresh milk was used as eye drop ( not exceed 6 hours after milking).
  Interventions: Biological: Breast milk
- Placebo group (Placebo Comparator): With in 48-72 hour after birth, infants will receive 0.5 ml 0.9% normal saline as a eye drop twice in a day until the discharge or need for laser coagulation.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Normal Saline — 0.5 ml 0.9% normal saline will drop on both eyes twice in a day.
  Arms: Placebo group
Biological: Breast milk — 0.5 ml breast milk from all infant's own mother will drop both eyes twice in a day
  Arms: Intervention group

SUMMARY:
The aim of this study is to investigate the effect of using breast milk as eye drops on ROP (Retinopathy of prematurity) disease observed in less then 32 weeks gestational age preterm babies.

DETAILED DESCRIPTION:
Study Design: Prospective randomized placebo controlled trial Setting/Participants: Premature babies who are at high risk for retinopathy of prematurity (ROP) during their stay in the neonatal intensive care unit (NICU). The study will be carried out at Baskent University and it is planned that 70 participants will be included in the study.

Study Interventions and Measures: After the randomization of the patients, 0.5 ml breast milk of the babies' own mothers will drop on the eye to the intervention group twice a day. IN the control group, %0.9 normal saline will drop as same amount. Primary outcome is any stage of ROP, secondary outcome is severe ROP (laser requiring ROP).

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 22 and 32 gestational age weeks or under 1500 gr birth weight.

Exclusion Criteria:

* Infant death before first examination for ROP
* parents who want to leave from the study
* Contraindications for breast milk use (Active HIV infection, Active tuberculosis, CMV infection)
* Inborn error of metabolism like galactosemia.
* Congenital eye development disorders like agenesis, or situations that do not allow retina examination.
* other lethal congenital molformations
* congenital infections that affect the retina like TORCH infections.

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Retinopathy of Prematurity | by 55 weeks post menstrual age
  Number of participants with any stage of ROP

SECONDARY OUTCOMES:
Retinopathy of Prematurity | by 55 weeks post menstrual age
  Number of participants with laser requiring - severe ROP

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No